CLINICAL TRIAL: NCT04455789
Title: Mechanical Ventilation in Lateral Position During Total Hip Replacement Surgery : Comparison of Driving Pressure With Conventional Ventilation
Brief Title: Mechanical Ventilation Based on Driving Pressure in Lateral Position
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: monitoring equipment used in the study is not available
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Nesil Coskunfirat, associate professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AkdenizU-2
Record Dates: First submitted 2020-06-25; First posted 2020-07-02 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Fracture of Hip; Osteoarthritis, Hip; Congenital Hip Deformity
Keywords: Driving Pressure; lung protective ventilation; PEEP; total hip replacement; lateral position
MeSH Terms: conditions — Hip Fractures; Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional mechanical ventilation (Experimental): routine mechanical ventilation will be adjusted based on conventional mechanical ventilation settings with tidal volume of 8 ml/kg and PEEP level of 5
  Interventions: Procedure: routine lung protective, conventional mechanical ventilation
- mechanical ventilation adjusted according to driving pressure (Experimental): routine mechanical ventilation adjusted based on driving pressure during lateral position. After patients are put to lateral position incremental increase in PEEP will be applied and the driving pressures will be recorded for each PEEP level and the patients will be ventilated with this PEEP during anesthesia. the other setting will be same with conventional group. tidal volume of 8 ml/kg
  Interventions: Procedure: routine lung protective, conventional mechanical ventilation

INTERVENTIONS:
Procedure: routine lung protective, conventional mechanical ventilation — routine lung protective, conventional mechanical ventilation with stabil PEEP
  Other Names: routine lung protective, conventional mechanical ventilation with PEEP adjusted to the lowest Driving Pressure level

SUMMARY:
Previous studies showed that, best lung protective strategies of ventilation parameters are based on driving pressure in damaged lungs. But there are few studies concerning the effects of different positions during different types of surgery on driving pressure with normal lungs.So the investigators decided to compare mechanical ventilation based on driving pressure with conventional mechanical ventilation in patients with lateral decubitus position during total hip replacement surgery. The investigators hypothesised that, there will be better intraoperative hemodynamic and respiratory parameters with better early postoperative results in patients whom mechanical ventilation parameters are adjusted according to driving pressure.

In this randomised, controlled, double blind study, 60 patients who will have total hip replacement surgery will be recruited to the study. 30 patients will be ventilated by 8 ml/kg tidal volume and 5 cmH20 PEEP, in conventional lung protective group. And the other 30 patients will be ventilated by 8 ml/kg tidal volume and PEEP level with the lowest driving pressure.

The investigators primary goal in this study study is to compare the effects of conventional lung protective ventilation with ventilation based on driving pressure on hemodynamic and respiratory parameters. And secondly, the investigators aim to compare the effects of these two techniques s on early postoperative outcome. The investigators primary result parameters are intra operative fluid consumption, lactate, etC02 and mix venous oxygen saturation levels.The investigators secondary result parameters are postoperative mechanical ventilation, ICU stay and discharge times.

DETAILED DESCRIPTION:
There may be physiologic and pathologic pulmonary changes because of inflammatory cytokine release during total hip replacement surgery due to surgical invasivity or advanced age, comorbidities, perioperative immobility of patients. Also intraoperative mechanical ventilation can cause volutrauma, barotrauma or atelectrauma risk because of lateral position during hip replacement surgery. All these factors can cause pulmonary complications and vascular permeability increase in dependent and independent regions due to neutrophil response increase. Intraoperative hypovolemia is often observed in this group patients because of preoperative prolonged fasting periods, insufficient fluid intake due to preoperative delirium and depression. Also mechanical ventilation with positive pressure slightly decreases venous return to the heart resulting decrease in cardiac output. It is more obvious in the presence of hypovolemia. Providing continuous sufficient intravascular volume is necessary for prevention of tissue hypoxia and providing optimal cardiac output. It is known that intra operative hemodynamic optimisation, has positive effects on mortality ratio. But proper intravascular volume is not always easy to maintain, and it is not always easy for anaesthetists to identify deficiency or overload of intra operative intravascular volume. In recent years, intravascular volume therapies are goal directed by the reflections of respiratory mechanics on arterial pressure and pulse oximetry. Plethysmographic wave changes observed in pulse oximetry induced by positive pressure ventilation is accepted as indicator of hypovolemia. Hemodynamic changes induced by respiratory mode can be measured by invasive arterial monitorization. This dynamic variable is called as pulse pressure variation index and is correlated with amplitude changes observed in pulse oximetry signals. These variations are based on changes observed in pulse wavelength due to the changes in intrathoracic pressure. In some pulse oximetry devices, this is done as standard function as path variability index (PVI). PVI is measurement of dynamic changes of perfusion index during a whole respiratory cycle. Pulse oximetry wave length changes enables the evaluate hypovolemia noninvasively.

PVI is gaining importance as a dynamic parameter in evaluating fluid treatment during surgery. Goal directed fluid therapy has shown positive effects on results on patient survival. In a study which fluid therapy was guided by PVI changes and it was reported that, goal directed fluid therapy had positive results.The investigators also, use some invasive and noninvasive monitorization techniques, including PVI and CVP, to monitor static and dynamic hemodynamic parameters during hip replacement surgery and we apply fluids according to our fluid therapy protocols. The investigators use blood gas analysis to monitor the efficiency of this treatment.

In this study, in both groups the investigators will apply fluid according to PVI values, so if any difference detected is observed between groups will be because of the differences of respiratory parameters between groups. And the investigators can detect, PVI stability and less fluid needs differences between groups.

PETCO2 is, another parameter which will be evaluated in this study, is a factor of tissue CO2 production (VCO2), alveolar ventilation and cardiac output (mainly pulmonary blood flow). It is known that, when CO2 produced at the tissues and formed in lungs are constant, the changes of etCO2 are due to the blood flow differences and it is related to changes of cardiac output. For this reason, PETCO2 is suggested as a noninvasive measure for continuous assessment of cardiac output. At the same time, it is possible to comment about changes of dead space by measuring arterial CO2 pressure.

Decrease of PETCO2, resulted from cardiac output decrease, can not be explained only with the decrease rate of excretion of CO2, but also can be explained by the changes of production of CO2 caused by dependency to oxygen supply. On the contrary, when cardiac output is high, pulmonary blood flow is no longer a limiting factor for PETCO2 formation, and PETCO2 is related to sufficiency of alveolar ventilation.

As a result, etCO2 measurement has some advantages; it is simple noninvasive and does not require a invasive hemodynamic measurement.

ELIGIBILITY:
Inclusion Criteria:

Patients planned to have total hip replacement

Exclusion Criteria:

High intracranial pressure Bronchopleural fistula Hypovolemic shock Right ventricular failure Left ventricular failure(Ejection fraction lower than 50%) Arrythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
volume of intraoperative fluid administration | during intraoperative period
  the patients will receive intraoperative fluids according to a protocol based on PVI.
intraoperative etCO2 levels | during mechanical ventilation
  et CO2 levels will be recorded form the anesthesia machine monitor
lactate levels | during intraoperative period
  lactate levels will be obtained from the serial blood gas analysis

SECONDARY OUTCOMES:
postoperative mechanical ventilation duration | From end of surgery to the end of mechanical ventilation duration in the intensive care unit until the patient is extubated, up to 3 days
  The patient's need for mechanical ventilation, after the surgery, will be assessed
postoperative intensive care stay | From end of operation to the end of intensive care stay, up to 1 week
  after the end of surgery the patients need for intensive care will be assessed
length of hospital stay after the operation | form end of surgery to the end of hospital stay, up to 10 days
  the effects of mechanical ventilation on the days of hospital stay will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye Bigat, Prof, Principal Investigator — Akdeniz University Medical School Anesthesiology and Reanimation Department; İlker O Aycan, Ass Prof, Principal Investigator — Akdeniz University Medical school Anesthesiology and Reanimation Departmnet
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No